CLINICAL TRIAL: NCT03091309
Title: Counseling to Optimize Medication Adherence in Expectant Mothers With Inflammatory Bowel Disease (COACH-IBD)
Brief Title: Counseling to Optimize Adherence in Expectant Mothers With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Crohn's and Colitis Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COACH-IBD
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Inflammatory Bowel Diseases; Medication Adherence; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Diseases; Medication Adherence; Crohn Disease; Ulcerative Colitis; Pregnancy; Counselling; Patient Education
MeSH Terms: conditions — Inflammatory Bowel Diseases; Medication Adherence; Crohn Disease; Colitis, Ulcerative | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to the intervention group will receive a multi-faceted intervention consisting of: (1) Interactive educational video; (2) Initial in-person counseling with an IBD nurse; (3) Motivational interviewing; (4) Telemedicine-based follow-up; (5) Monthly follow-up questionnaires; and (6) Comprehensive questionnaires.
  Interventions: Other: Interactive educational video; Behavioral: Initial in-person counseling with an IBD nurse; Behavioral: Motivational interviewing; Behavioral: Telemedicine-based follow-up; Other: Monthly follow-up questionnaires; Other: Comprehensive questionnaires
- Control (Active Comparator): Patients randomized to the control group will complete the comprehensive questionnaires and will continue to receive the standard of care consistent with their condition, at their respective institution.
  Interventions: Other: Comprehensive questionnaires

INTERVENTIONS:
Other: Interactive educational video — A web-link to an educational video on IBD and pregnancy tailored to emphasize the importance of optimal disease control and medication adherence.
  Arms: Intervention
Behavioral: Initial in-person counseling with an IBD nurse — This session will emphasize key points from the educational video and the nurse will answer any additional questions the subject may have. The nurse will assess subjects' medication adherence and specifically query any concerns subjects may have regarding specific medications and discuss their intentions to be adherent throughout pregnancy.
  Arms: Intervention
Behavioral: Motivational interviewing — The nurse will be trained in a technique known as motivational interviewing (MI) specifically adapted for optimizing medication adherence during pregnancy.
  Arms: Intervention
Behavioral: Telemedicine-based follow-up — The IBD nurse will arrange follow-up visits with each subject on a monthly basis with additional ad-hoc sessions as needed. The encounter will focus on monitoring disease activity adherence and applying MI communication skills to reinforce and improve the latter.
  Arms: Intervention
Other: Monthly follow-up questionnaires — Web-based short questionnaires, administered monthly, will be used to assess medication adherence [self-reported using the 5 item Medication Adherence Report Scale (MARS-5)] and IBD related disease activated [self-reported using PRO-2 scale for Crohn's Disease related disease activity and 6-Point Mayo Score for Ulcerative Colitis related disease activity].
  Arms: Intervention
Other: Comprehensive questionnaires — Web-based detailed questionnaires, administered at enrolment and gestational week 34, will be used to assess medication adherence [self-reported using the Medication Adherence Report Scale (MARS-5)], patient trust in physician [self-reported using the Trust in Physician Scale (TIPS)], IBD related disease activated [self-reported using the PRO-2 or 6-Point Mayo Score], IBD-specific health related quality of life [self-reported using the Inflammatory Bowel Disease Questionnaire (IBDQ)], patient satisfaction [self-reported using the Patient Satisfaction with Healthcare in Inflammatory Bowel Disease (CACHE) questionnaire]and IBD specific knowledge [self-reported using the Crohn's and Colitis Knowledge (CCKNOW) questionnaire].

SUMMARY:
Inflammatory Bowel Disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract that comprises two subtypes, Crohn's disease (CD) and Ulcerative Colitis (UC). Because the risk of IBD is greatest during the third decade of life, its impact for women is during the reproductive years. Women with inflammatory bowel disease are at a 2-fold higher risk of adverse outcomes during pregnancy as compared to the general population. Pregnancy is an especially vulnerable time for women with IBD, and out of misguided concerns that medications may confer unnecessary harms to their fetus, many women often stop taking life savings medications; without realizing that this sub-optimal adherence could actually lead to life threatening complications for them and their fetus. Counseling pregnant women with IBD is therefore an important step in improving medication adherence. The investigators hypothesize that counseling sessions with an IBD nurse that incorporates motivational interviewing and telemedicine-based follow-up sessions tailored to individual needs will improve medication adherence and pregnancy outcomes.

The following specific aims are to be addressed by this multi-center randomized clinical trial comparing individual nurse-based counseling to standard of care:

Specific Aim #1: To assess whether patient-centered counseling incorporating motivational interviewing and telemedicine-based follow-up by an IBD nurse leads to improved medication adherence during pregnancy and pregnancy outcomes

Specific Aim #2: To validate the use of self-reported medication adherence during pregnancy in the IBD population

DETAILED DESCRIPTION:
IBD and Pregnancy: Inflammatory bowel disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract that comprises two subtypes, Crohn's disease (CD) and Ulcerative Colitis (UC), Canada has among the highest reported incidence of CD and UC in the world, as high as 20.2 and 19.5 per 100,000, respectively. Because the risk of IBD is greatest during the third decade of life, its greatest impact for women in during the reproductive years. In comparison to the general population, women with IBD have a significantly higher risk of pregnancy related complications.

IBD Disease Activity and Outcomes: Active IBD symptoms during pregnancy significantly increase the risk of preterm birth. Furthermore, women with IBD who suffer a relapse during pregnancy, requiring hospitalization, are more likely than their asymptomatic counterparts to delivery preterm birth and low birth weight newborns. More than two-thirds of women who have active disease at the time of conception will have continued or worsened symptoms during pregnancy. In contrast, women who are asymptomatic at conception are half as likely to have active disease during pregnancy. This data underscores the importance of achieving disease remission prior to conception and aggressively treating relapses during pregnancy.

Medication Adherence During Pregnancy: Despite the safety of most IBD medications, most pregnant women with IBD exhibit low medication adherence rates. Medication non-compliance is often linked to concerns that IBD medication may confer unnecessary harm to the fetus. Most women have reported that they would rather endure symptoms of IBD rather than confer risk to the fetus, without realizing that active IBD itself is strongly associated with adverse pregnancy outcomes. Consequently, most of these women decrease the dosage or stop their medications without informing their treating physicians, thus comprising treatment.

Motivational Interviewing Adherence: Motivational Interviewing (MI) refers to a patient-centered process in which a health care provider employs specific communication skills and strategies that facilitate the patients confidence and decision making, while emphasising respect for autonomy. A key feature of MI is that the counselling process induces behavioural change by triggering and channelling a patient's internal motivations for change. Previous clinical trials have demonstrated the effectiveness of MI in improving medication adherence for various chronic condition, including diabetes, hypertension, obesity and HIV. In a small study of IBD subjects, MI was associated with positive patient perceptions of the physician-patient relationship. In another pilot study, nurse-administered MI in UC patients was associated with medication adherence as high as 90%.

Rationale: Pregnancy is an especially vulnerable time for women with IBD. During this critical window of time, even brief lapses in medication adherence can lead to sub optimal control of IBD disease activity that can lead to life-threatening complications to both mother and fetus. Adverse outcomes such as preterm delivery have long-term implications for the children of mother with IBD. Out of misguided concerns for their fetus, many women may stop lifesaving medications. Educating pregnant women with IBD is an important step in improving adherence rates, but tools such as motivational interviewing have proven to be much more powerful. As such the primary objective of this study is to assess, through a multi-center clinical trial, whether patient-centered counselling incorporating motivational interviewing and telemedicine-based follow-up by an IBD nurse leads to improved medication adherence during pregnancy and improved pregnancy outcomes. The investigators hypothesize that patient-centered counselling will result in higher medication adherence rates and improved pregnancy outcomes.

Design: The investigators will conduct a multi-center randomized controlled clinical trial that includes 3 University of Toronto affiliated hospitals (Mount Sinai Hospital, University Health Network, and Women's College Hospital) and the University of Calgary.

Study Population: The investigators will enroll 220 pregnant women who have or will be seen by: an obstetrician or maternal fetal specialist at Mount Sinai Hospital or the University of Calgary; or a gastroenterologist at Mount Sinai Hospital, University Health Network, Women's College, or the University of Calgary who meet the inclusion criteria.

Significance: This clinical intervention has the potential to directly impact inflammatory bowel disease patients by reducing complications of the disease during pregnancy. Motivational interviewing can potentially improve adherence and optimize the impact of IBD medical therapies. Most tertiary centers already have clinical IBD nurses. The structured training of an IBD nurse to counsel pregnant women through motivational interviewing is a reproducible intervention and can be used at tertiary centers throughout the country. Because poor disease control can lead to preterm delivery, which is associated with lifelong chronic illnesses, patient-centered counselling would not only ameliorate the IBD health of mothers, but also improve the lives of their children. Findings from this study would also allow physicians to lobby provincial health ministries to request funds for IBD nurse counsellors.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of IBD
* Expected to be on an IBD-related medication throughout pregnancy
* In First Trimester of Pregnancy
* Willing to undergo pregnancy counseling with close monitoring
* Able to provide informed consent

Exclusion Criteria:

* Patients who are not residing in Ontario of Alberta
* Unconfirmed diagnosis of IBD
* In Second or Third Trimester of Pregnancy
* Uncertainty regarding whether IBD medication will be prescribed throughout pregnancy
* Unwilling to participate
* Inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 220 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence (MARS-5) | Comparison of dichotomous variable at Baseline and Gestational Week 34
  Comparison of medication adherence as a dichotomous outcome (adherent vs. non-adherent) using the chi-square statistic between intervention and control groups.

SECONDARY OUTCOMES:
IBD-Specific Health Related Quality of Life (IBDQ) | Comparison of continuous variable at Baseline Gestational Week 34
  Comparison of IBDQ as a continuous variable using the the Mann-Whitney test between intervention and control groups.
PRO-2 Scale for Crohn's Disease related disease activity | Comparison of continuous variable at Baseline Gestational Week 34
  Comparison of scores on the PRO-2 scores as a continuous variable using the the Mann-Whitney test between intervention and control groups.
6-Point Mayo Score for Ulcerative Colitis related disease activity | Comparison of continuous variable at Baseline Gestational Week 34
  Comparison of 6-Point Mayo Score as a continuous variable using the the Mann-Whitney test between intervention and control groups.
Patient Trust in Physician (TIPS) | Comparison of continuous variable at Baseline Gestational Week 34
  Comparison of TIPS as a continuous variable using the the Mann-Whitney test between intervention and control groups.
Patient Satisfaction (CACHE) | Comparison of continuous variable at Baseline Gestational Week 34
  Comparison of CACHE as a continuous variable using the the Mann-Whitney test between intervention and control groups.
IBD Specific Knowledge (CCKNOW) | Comparison of continuous variable at Baseline Gestational Week 34
  Comparison of CCKNOW as a continuous variable using the the Mann-Whitney test between intervention and control groups.
Fecal Calprotectin | Comparison of dichotomous outcome at Baseline and Gestational Week 34
  Comparison of proportion of subjects with elevated fecal calprotectin scores, as an objective measure of inflammation and disease activity, between study groups using chi-square statistic.
Preterm Delivery | Comparison of dichotomous outcome at Delivery
  Gestational age recorded at delivery will be used to ascertain preterm delivery (<37 weeks) and compare rates of preterm delivery between study groups using chi-square statistic.
Small for Gestational Age | Comparison of dichotomous outcome at Delivery
  Birth weight recorded at delivery will be used to ascertain whether infants are small for gestational age and compare rates of small for gestational age infants at delivery between study groups using chi-square statistic.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Nguyen, MD, PhD, Principal Investigator — Mount Sinai Hospital (Toronto, ON, Canada)
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norgard B, Hundborg HH, Jacobsen BA, Nielsen GL, Fonager K. Disease activity in pregnant women with Crohn's disease and birth outcomes: a regional Danish cohort study. Am J Gastroenterol. 2007 Sep;102(9):1947-54. doi: 10.1111/j.1572-0241.2007.01355.x. Epub 2007 Jun 15. PMID 17573787
- [Background] Reddy D, Murphy SJ, Kane SV, Present DH, Kornbluth AA. Relapses of inflammatory bowel disease during pregnancy: in-hospital management and birth outcomes. Am J Gastroenterol. 2008 May;103(5):1203-9. doi: 10.1111/j.1572-0241.2007.01756.x. Epub 2008 Apr 16. PMID 18422816
- [Background] Abhyankar A, Ham M, Moss AC. Meta-analysis: the impact of disease activity at conception on disease activity during pregnancy in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2013 Sep;38(5):460-6. doi: 10.1111/apt.12417. Epub 2013 Jul 15. PMID 23855477
- [Background] Selinger CP, Eaden J, Selby W, Jones DB, Katelaris P, Chapman G, McDondald C, McLaughlin J, Leong RW, Lal S. Inflammatory bowel disease and pregnancy: lack of knowledge is associated with negative views. J Crohns Colitis. 2013 Jul;7(6):e206-13. doi: 10.1016/j.crohns.2012.09.010. Epub 2012 Oct 2. PMID 23040449
- [Background] Mountifield RE, Prosser R, Bampton P, Muller K, Andrews JM. Pregnancy and IBD treatment: this challenging interplay from a patients' perspective. J Crohns Colitis. 2010 Jun;4(2):176-82. doi: 10.1016/j.crohns.2009.10.001. Epub 2009 Dec 4. PMID 21122502
- [Background] Fidder HH, Singendonk MM, van der Have M, Oldenburg B, van Oijen MG. Low rates of adherence for tumor necrosis factor-alpha inhibitors in Crohn's disease and rheumatoid arthritis: results of a systematic review. World J Gastroenterol. 2013 Jul 21;19(27):4344-50. doi: 10.3748/wjg.v19.i27.4344. PMID 23885145
- [Background] Britt E, Hudson SM, Blampied NM. Motivational interviewing in health settings: a review. Patient Educ Couns. 2004 May;53(2):147-55. doi: 10.1016/S0738-3991(03)00141-1. PMID 15140454
- [Background] Easthall C, Song F, Bhattacharya D. A meta-analysis of cognitive-based behaviour change techniques as interventions to improve medication adherence. BMJ Open. 2013 Aug 9;3(8):e002749. doi: 10.1136/bmjopen-2013-002749. PMID 23935093
- [Background] Hedegaard U, Kjeldsen LJ, Pottegard A, Henriksen JE, Lambrechtsen J, Hangaard J, Hallas J. Improving Medication Adherence in Patients with Hypertension: A Randomized Trial. Am J Med. 2015 Dec;128(12):1351-61. doi: 10.1016/j.amjmed.2015.08.011. Epub 2015 Aug 21. PMID 26302142
- [Background] Ekong G, Kavookjian J. Motivational interviewing and outcomes in adults with type 2 diabetes: A systematic review. Patient Educ Couns. 2016 Jun;99(6):944-52. doi: 10.1016/j.pec.2015.11.022. Epub 2015 Dec 4. PMID 26699083
- [Background] Barnes RD, Ivezaj V. A systematic review of motivational interviewing for weight loss among adults in primary care. Obes Rev. 2015 Apr;16(4):304-18. doi: 10.1111/obr.12264. Epub 2015 Mar 5. PMID 25752449
- [Background] Armstrong MJ, Mottershead TA, Ronksley PE, Sigal RJ, Campbell TS, Hemmelgarn BR. Motivational interviewing to improve weight loss in overweight and/or obese patients: a systematic review and meta-analysis of randomized controlled trials. Obes Rev. 2011 Sep;12(9):709-23. doi: 10.1111/j.1467-789X.2011.00892.x. Epub 2011 Jun 21. PMID 21692966
- [Background] Hill S, Kavookjian J. Motivational interviewing as a behavioral intervention to increase HAART adherence in patients who are HIV-positive: a systematic review of the literature. AIDS Care. 2012;24(5):583-92. doi: 10.1080/09540121.2011.630354. Epub 2012 Jan 31. PMID 22292452
- [Background] Mocciaro F, Di Mitri R, Russo G, Leone S, Quercia V. Motivational interviewing in inflammatory bowel disease patients: a useful tool for outpatient counselling. Dig Liver Dis. 2014 Oct;46(10):893-7. doi: 10.1016/j.dld.2014.07.009. Epub 2014 Jul 30. PMID 25085685
- [Background] Cook PF, Emiliozzi S, El-Hajj D, McCabe MM. Telephone nurse counseling for medication adherence in ulcerative colitis: a preliminary study. Patient Educ Couns. 2010 Nov;81(2):182-6. doi: 10.1016/j.pec.2009.12.010. Epub 2010 Jan 15. PMID 20079598
- [Background] Saghaei M. An overview of randomization and minimization programs for randomized clinical trials. J Med Signals Sens. 2011 Jan;1(1):55-61. PMID 22606659
- [Background] Trindade AJ, Ehrlich A, Kornbluth A, Ullman TA. Are your patients taking their medicine? Validation of a new adherence scale in patients with inflammatory bowel disease and comparison with physician perception of adherence. Inflamm Bowel Dis. 2011 Feb;17(2):599-604. doi: 10.1002/ibd.21310. PMID 20848512
- [Background] Rocchi A, Benchimol EI, Bernstein CN, Bitton A, Feagan B, Panaccione R, Glasgow KW, Fernandes A, Ghosh S. Inflammatory bowel disease: a Canadian burden of illness review. Can J Gastroenterol. 2012 Nov;26(11):811-7. doi: 10.1155/2012/984575. PMID 23166905
- [Background] Bernstein CN, Wajda A, Svenson LW, MacKenzie A, Koehoorn M, Jackson M, Fedorak R, Israel D, Blanchard JF. The epidemiology of inflammatory bowel disease in Canada: a population-based study. Am J Gastroenterol. 2006 Jul;101(7):1559-68. doi: 10.1111/j.1572-0241.2006.00603.x. PMID 16863561
- [Background] Cornish J, Tan E, Teare J, Teoh TG, Rai R, Clark SK, Tekkis PP. A meta-analysis on the influence of inflammatory bowel disease on pregnancy. Gut. 2007 Jun;56(6):830-7. doi: 10.1136/gut.2006.108324. Epub 2006 Dec 21. PMID 17185356
- [Background] Dominitz JA, Young JC, Boyko EJ. Outcomes of infants born to mothers with inflammatory bowel disease: a population-based cohort study. Am J Gastroenterol. 2002 Mar;97(3):641-8. doi: 10.1111/j.1572-0241.2002.05543.x. PMID 11926208
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391